CLINICAL TRIAL: NCT03369197
Title: A Randomized Controlled Trial of an Intervention to Reduce the Incidence of Hypoxia With Nasal Continuous Positive Airway Pressure Versus Standard Care During Procedural Sedation for Gastrointestinal Endoscopy
Brief Title: Nasal Continuous Positive Airway Pressure Versus Standard Care During Procedural Sedation for Gastrointestinal Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00118466
Record Dates: First submitted 2017-11-28; First posted 2017-12-11 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Hypoxia; Endoscopy; Anesthesia Morbidity
Keywords: procedural sedation; monitored anesthesia care; endoscopy
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention: Nasal Mask (Experimental): Nasal anesthesia mask with positive pressure
  Interventions: Device: Nasal Mask
- Control: Nasal cannula (Active Comparator): Nasal Cannula with standard care
  Interventions: Device: Control: Nasal Cannula

INTERVENTIONS:
Device: Nasal Mask — Nasal anesthesia mask which covers the nose and attaches to the anesthesia circuit, allowing for variable positive pressure by setting the pop-off valve
  Other Names: Intervention: Nasal anesthesia mask with positive pressure
  Arms: Intervention: Nasal Mask
Device: Control: Nasal Cannula — Nasal cannula as per usual care
  Other Names: Standard Care
  Arms: Control: Nasal cannula

SUMMARY:
This study is a randomized controlled trial comparing oxygen delivery by nasal mask with continuous positive airway pressure versus standard care (nasal cannula or standard facemask) during propofol-based sedation for gastrointestinal endoscopy procedures to reduce the incidence of hypoxia. The primary outcome will be the rate of oxygen desaturation below 90% for ≥15 seconds.

DETAILED DESCRIPTION:
This study is a randomized controlled trial comparing oxygen delivery by nasal mask with continuous positive airway pressure versus standard care (nasal cannula or standard facemask) during propofol-based sedation for gastrointestinal endoscopy procedures to reduce the incidence of hypoxia. The primary outcome will be the rate of oxygen desaturation below 90% for ≥15 seconds. In addition, secondary measures will include evaluation of mechanism and degree of respiratory depression associated with hypoxia and hypoventilation by characterizing changes in minute ventilation, tidal volume, and respiratory rate as well as the rate and degree of airway obstruction. The investigators hypothesize that the addition of nasal continuous positive airway pressure in the intervention arm will lead to decreased obstruction as positive pressure will stent open the obstructed airway. Depth of anesthesia will be monitored by Bispectral Index and investigators hypothesize that the degree of hypoventilation, obstruction, and will be significantly lower in the intervention arm compared to the control arm. Further, the depth of anesthesia will be independent of total propofol dose received. While the primary outcome in this study is hypoxia, investigators also seek to marry end tidal carbon dioxide with minute ventilation and transcutaneous carbon dioxide measurement to better understand the total effects of sedation on respiration. Thus the study will also serve to evaluate which mode(s) of respiratory monitoring might be the best possible intervention to enhance safety during procedural sedation in the future. Further, investigators suspect that the amplitude of end tidal carbon dioxide will not predict the degree of respiratory depression seen with other monitors. In addition, investigators will measure serum short chain fatty acid concentrations as a predictor and possible mechanism for differences in individual variability in anesthesia induced respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age) undergoing colonoscopy, endoscopic gastroduodenoscopy, and endoscopic gastroduodenoscopy with biopsy and/or ultrasound, or combined upper and lower endoscopy procedure anticipated to last longer than 10 minutes in the Endoscopy Suite at the Johns Hopkins Hospital when the anesthetic plan is monitored anesthesia care with propofol-based anesthesia with a natural airway.

Exclusion Criteria:

* Left ventricular Assist Device
* Severe Pulmonary Hypertension
* Ejection fraction less than 35 percent
* Active Congestive Heart Failure Exacerbation
* Planned procedure is Balloon Enteroscopy or Endoscopic Retrograde Duodenoscopy.
* Topical lidocaine administration
* Pregnancy
* Previous enrollment in this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laeben Lester, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the Endoscopy suite at Johns Hopkins Hospital.
Period: Overall Study
Arm/Group | Intervention: Nasal Mask | Control: Nasal Cannula
Started | 53 | 58
Completed | 53 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: Nasal Mask | Control: Nasal Cannula | Total
Number analyzed (Participants) | 53 | 58 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 42 | 72
  >=65 years | 23 | 16 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 29 | 29 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 53 | 57 | 110
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 12 | 19
  White | 42 | 44 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Hypoxia Rate as Assessed by Number of Participants With at Least One Hypoxic Event
Description: Number of subjects undergoing procedural sedation for endoscopy with at least one hypoxic event, defined as oxygen saturation less than 90 percent for 15 seconds.
Time Frame: Approximately 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Nasal Mask | Control: Nasal Cannula
Number analyzed (Participants) | 53 | 58
Participants | 3 | 16

2. Secondary Outcome: Hypoventilation in Subjects Undergoing Procedural Sedation for Endoscopy as Assessed by Transcutaneous Carbon Dioxide Monitoring
Description: Evaluate hypoventilation in subjects undergoing procedural sedation for endoscopy by transcutaneous carbon dioxide monitoring in millimeters of mercury (mmHg).
Time Frame: Approximately 1 hour
Population: 11 participants from intervention group and 9 participants from control group were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention: Nasal Mask | Control: Nasal Cannula
Number analyzed (Participants) | 42 | 48
mmHg | 53.3 (6.20) | 51.9 (8.14)

3. Secondary Outcome: Hypoventilation in Subjects Undergoing Procedural Sedation for Endoscopy as Assessed by Respiratory Volume Monitoring
Description: Evaluate hypoventilation by respiratory volume monitoring for minute ventilation. Reported result is the percentage decrease from baseline in minute ventilation.
Time Frame: Approximately 1 hour
Population: Only 43 in the intervention group and 40 in the control group had sufficient data to be analyzed.
Measure: Mean (Standard Deviation); unit: percentage of decrease
Arm/Group | Intervention: Nasal Mask | Control: Nasal Cannula
Number analyzed (Participants) | 43 | 40
percentage of decrease | 64 (21.9) | 59 (22)

4. Secondary Outcome: Mechanism of Hypoventilation in Subjects Undergoing Procedural Sedation for Endoscopy and Hypoventilation
Description: Correlate respiratory volume monitoring transcutaneous carbon dioxide measurement with number of airway maneuvers to identify mechanism of hypoventilation as predominately obstructive or due to respiratory rate or tidal volume.
Time Frame: Approximately 1 hour
Population: This data was not collected.
Arm/Group | Intervention: Nasal Mask | Control: Nasal Cannula
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Depth of Anesthesia in Subjects Undergoing Procedural Sedation for Endoscopy
Description: Depth of anesthesia by processed electroencephalogram (EEG) bispectral analysis, which is a standard monitor of anesthetic depth using a calibrated dimensionless index that ranges from 0 to 100, with lower numbers corresponding to a deeper anesthetic state.
Time Frame: Approximately 1 hour
Population: 5 participants from intervention group and 7 participants from control group were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Nasal Mask | Control: Nasal Cannula
Number analyzed (Participants) | 48 | 50
score on a scale | 40.19 (13.64) | 40.30 (15.07)

6. Secondary Outcome: Hypoxia Duration
Description: The total time in seconds of oxygen saturation below 90 percent will be recorded
Time Frame: Approximately 1 hour
Population: This data was not collected.
Arm/Group | Intervention: Nasal Mask | Control: Nasal Cannula
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Total Number of Hypoxic Events in Subjects That Experienced Hypoxia
Description: In subjects experiencing hypoxia during sedation, the total number of episodes of hypoxia for all participants will be recorded.
Time Frame: Approximately 1 hour
Population: The 3 patients in nasal mask arm and 16 in nasal cannula arm experienced hypoxia.
Measure: Number; unit: hypoxic events
Arm/Group | Intervention: Nasal Mask | Control: Nasal Cannula
Number analyzed (Participants) | 3 | 16
hypoxic events | 4 | 23

8. Other Pre Specified Outcome: Short Chain Fatty Acid Concentration
Description: Measure baseline short chain fatty acids in subjects undergoing procedural sedation for endoscopy and correlate the concentration with the degree of respiratory depression by respiratory volume monitoring and transcutaneous carbon dioxide.
Time Frame: Approximately 1 hour
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Discharge from endoscopy unit, up to 1 week.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Intervention: Nasal Mask | Control: Nasal Cannula
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/57
Other Adverse Events (participants affected / at risk) | 0/53 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT03369197/Prot_SAP_001.pdf
  • Informed Consent Form (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT03369197/ICF_000.pdf